CLINICAL TRIAL: NCT03742648
Title: The Effectiveness of Deep Breathing Exercises in Second Degree Inhalational Burns
Brief Title: The Effectiveness of Deep Breathing Exercises and Incentive Spirometry in Second Degree Inhalation Burn Patients
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isra University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1502-PDPT-005
Record Dates: First submitted 2018-10-25; First posted 2018-11-15 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Burn Patients
Keywords: pO2; pCO2; pH; Rhonchi; Wheeze; Crackles; ISM; DBE
MeSH Terms: conditions — Respiratory Sounds | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two or more groups in parallel for the duration of the study
Masking Description: There is no party who is masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control physiotherapy group (Active Comparator): Basic standard medical and nursing care along with standard chest physiotherapy involving steam inhalation and nebulization for 15-20 minutes and 10-15 cycles of incentive spirometry twice daily
  Interventions: Other: Physiotherapy
- Experimental physiotherapy group (Experimental): Basic standard medical and nursing care along with chest physiotherapy involving any of the deep breathing exercises as per patients ease with 5-10 repetitions each, twice daily
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy — Chest physiotherapy in burn patients in order to treat and prevent post burn respiratory complications like pneumonia etc
  Other Names: Chest physiotherapy

SUMMARY:
The purpose of the study was to find out the effectiveness of the Deep Breathing Exercises and Incentive Spirometry in Second degree inhalation Burn patients and to find out best effective method.It was a Randomized Control Trial performed on the patients of Pakistan Institute of Management Sciences hospital Islamabad for duration of 06 months after approval of synopsis.30 patients of second degree inhalation burns between the age of 20-50 years having good pre burn respiratory state and irrespective of gender discrimination who were currently on nasal cannula were randomly allocated in control and experimental groups.However all unconscious patients other than second degree inhalation burn and having comorbidities were excluded. The conventional treatment with steam inhalation and nebulization followed by Incentive spirometry with 10-15cycles and the treatment session lasts for 35-45 minutes for a period of 07 days with two sessions of this protocol were given to control group each day.For experimental group patients were made to perform different types of deep breathing exercises with 5-10 repetitions for a period of 07days with two sessions of this treatment protocol each day. Self structured questionnaires with informed consents were used to assess the data on day 00 and day 07 by Physiotherapist.The data was then analyzed using SPSS version 21.0.The results were then formulated using statistical analysis and then were arranged in different tables and graphs.

DETAILED DESCRIPTION:
Objective: To find out the effectiveness of the Deep Breathing Exercises and Incentive Spirometry in Second degree inhalation Burn patients and to find out best effective method.

Study Design:It is a Randomized Control Trial. Place and Duration of Study: Data was collected from Department of Burn, Pakistan Institute of Management Sciences hospital Islamabad, the study duration is 06 months after approval of synopsis.

Methodology: A total of 30 Second degree inhalation burn patients were included. Inclusion criteria includes both genders of patients between the ages of 20 to 50 years,with good Pre-Burn respiratory state and currently on Nasal Cannula.They were then randomly allocated using lottery method in control and experimental groups. Exclusion criteria includes all unconscious patients other than second degree inhalation burn and with other comorbidities.The treatment protocol designed for control group involves conventional treatment with steam inhalation and nebulization followed by Incentive spirometry with 10-15 cycles,the treatment session lasts for 35-45 minutes for a period of 07 days with two sessions of this protocol each day.The treatment protocol for experimental group includes different types of deep breathing exercises with 5-10 repetitions for a period of 07days with two sessions of this treatment protocol each day.The data was collected through self-structured questionnaires containing 17 questions and each question has four options.Baseline data was collected on Day 00 and then on Day 07 data was recollected for comparison of both groups by Physiotherapist.

ELIGIBILITY:
Inclusion Criteria:

* All the patients suffering from Second Degree inhalation Burn.
* Both genders will be included with good Pre-Burn respiratory state.
* All the patients after first surgical intervention, using mask and nasal cannulas, between the age of 20 - 50 years.

Exclusion Criteria:

* Patients suffering from other types of burns e.g. chemical etc.
* All the unconscious patients/ventilator dependent patients.
* All the patients with co-morbidities including COPD, Emphysema.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Changes in values of Arterial Blood gases- pH | On day 01 and on day 07
  Standard values taken as pH= 7.34-7.35
Changes in values of Arterial Blood Gases-pO2 | On day 01 and on day 07
  Standard values taken as pO2= 88-100 mmHg
Changes in values of Arterial Blood Gases- pCO2 | On day 01 and on day 07
  Standard values taken as pCO2= 45-55 mmHg

SECONDARY OUTCOMES:
Changes in Respiratory distress score(lag=0,normal=1, lead=2) | On day 01 and on day 07
  Chest movement, Intercostal retractions, Xiphoid retractions, Nasal flaring, Expiratory grunt
Change in Chest status/auscultation | On day 01 and on day 07
  Wheeze, Rhonchi, Crackles
Change in Vital signs | On day 01 and on day 07
  Temperature
Change in Pulse rate | On day 01 and on day 07
  Pulse rate per minute
Change in Respiratory rate | On day 01 and on day 07
  Respiratory rate per minute
Change in Blood pressure | On day 01 and on day 07
  Blood pressure in mmHg
Change in SaO2 | On day 01 and on day 07
  Oxygen saturation in %

CONTACTS AND LOCATIONS:
Overall Officials: Waqar A Awan, PhD, Study Chair — Isra University Islamabad Campus
Locations (1):
- Summyia Siddique Malik, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
Can be shared purposefully

REFERENCES:
- [Result] Cox RA, Burke AS, Soejima K, Murakami K, Katahira J, Traber LD, Herndon DN, Schmalstieg FC, Traber DL, Hawkins HK. Airway obstruction in sheep with burn and smoke inhalation injuries. Am J Respir Cell Mol Biol. 2003 Sep;29(3 Pt 1):295-302. doi: 10.1165/rcmb.4860. PMID 12936906